CLINICAL TRIAL: NCT06663007
Title: Prospective, Single Arm, Multi Cohort Clinical Study of Disitamab Vedotin(RC48) Monotherapy or Combination With Envafolimab for Second-line Treatment of CDK12 Alterations Metastatic Castration Resistant Prostate Cancer With Standard Treatment Failure
Brief Title: RC48 Monotherapy or Combination With Envafolimab for CDK12 Alterations mCRPC With Standard Treatment Failure
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RC48-mCRPC
Record Dates: First submitted 2024-10-26; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer; CDK12 Gene Mutation
MeSH Terms: conditions — Prostatic Neoplasms | interventions — disitamab vedotin; envafolimab

STUDY DESIGN:
Intervention Model Description: Simon's two-stage design.If the number of valid cases in the first stage is less than or equal to 0, the study will be terminated prematurely. If the number of valid cases in the first stage is greater than 0, participants will continue to be enrolled in the second stage. If the total number of valid cases is greater than 3 after the completion of the second stage, the queue experimental group is considered valid.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): During the treatment phase of patients in cohort A (excluding CDK12 alterations from mutation spectrum features in cohort B), subjects received intravenous infusion of Disitamab Vedotin(RC48) (2.0 mg/kg) every 2 weeks, in combination with subcutaneous injection of Envafolimab (400 mg) every 3 weeks, until disease progression or death occurred.
  Interventions: Drug: RC48; Drug: Envafolimab
- Cohort B (Experimental): During the treatment phase, subjects in cohort B (CDK12 alterations combined with 11q13 co-amplification, MDM2/4 amplification, FGFRs amplification and other chromosomal unstable mutation profiles) received intravenous infusion of Disitamab Vedotin(RC48) (2.0 mg/kg) every 2 weeks until disease progression or death occurred.
  Interventions: Drug: RC48

INTERVENTIONS:
Drug: RC48 — During the patient treatment phase, the subjects received intravenous infusion of Disitamab Vedotin(RC48) (2.0 mg/kg) every 2 weeks until disease progression or death occurred.
  Other Names: Disitamab Vedotin
Drug: Envafolimab — During the treatment phase of the patient, the subjects received subcutaneous injections of Envafolimab (400 mg) every 3 weeks until the patient experienced disease progression or death.
  Arms: Cohort A

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of vediximab monotherapy or in combination with enrolizumab for second-line treatment of CDK12 alterations mCRPC that has failed standard therapy. The research results are expected to provide new insights and breakthroughs for the treatment of advanced prostate cancer.

DETAILED DESCRIPTION:
This study plans to enroll 72 mCRPC patients who have failed at least one NHT standard treatment and have exhausted PARPi treatment (such as AVPC/NEPC, requiring platinum chemotherapy resistance or intolerance). The patient carries CDK12 mutation combined with ERBB amplification (NGS or FISH) or HER2 IHC (1+, 2+, 3+). The enrolled patients were divided into queue A and queue B based on whether they carried potential immunotherapy adverse factors (including chromosome instability mutation profiles such as 11q13 co amplification, MDM2/4 amplification, FGFRs amplification, etc.). During the treatment phase of patients in queue A (excluding CDK12mut from mutation spectrum features in queue B), subjects received intravenous infusion of vediximab (2.0 mg/kg) every 2 weeks, in combination with subcutaneous injection of bevacizumab (400 mg) every 3 weeks, until disease progression or death occurred. During the treatment phase, subjects in queue B (CDK12mut combined with 11q13 co amplification, MDM2/4 amplification, FGFRs amplification and other chromosomal unstable mutation profiles) received intravenous infusion of vediximab (2.0 mg/kg) every 2 weeks until disease progression or death occurred. The main endpoint of the study was hierarchical testing, Step 1: ORR in CDK12 mut mCRPC with ERBB2 IHC 3+or FISH+or ERBB amplification (CN ≥ 4); Step2: ORR in ITT。 The secondary endpoints of the study include PSA50, PFS, OS, and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be able to understand the procedures and methods of this study, willing to strictly follow the clinical trial protocol to complete the trial, and voluntarily sign a written informed consent form;
2. Patients aged ≥ 18 years old;
3. Pathological examination confirms non resectable or metastatic HER2 positive castration resistant prostate cancer (mCRPC): HER2 positive is defined as IHC 3+or IHC 2+or FISH+;
4. Carrying CDK12 mutation combined with ERBB amplification (NGS or FISH) or HER2 IHC (1+, 2+, 3+);
5. According to the RECIST solid tumor efficacy evaluation criteria, there must be at least one measurable lesion;
6. ECOG PS: 0-2 points;
7. Expected survival period is not less than 12 weeks;
8. Prior exposure to at least one novel endocrine therapy (including abiraterone, enzalutamide, darotamine, apatamide, and rivalutamide) and depletion of PARPi treatment (if AVPC/NEPC, platinum chemotherapy resistance or intolerance is required);
9. Have not used HER2 targeted drugs (including antibodies, small molecule TKIs, and antibody drug conjugates);
10. The main organ functions are normal, which meets the following criteria:

1) The standard for blood routine examination should meet the requirement of: Hb ≥ 90g/L (no blood transfusion or blood products within 14 days, no correction with G-CSF or other hematopoietic stimulating factors); ANC≥1.5×109/L； PLT≥90×109/L； 2) Biochemical tests must meet the following standards: TBiL≤1×ULN； ALT and AST ≤ 1.5 × ULN; ALP≤2.5×ULN； BUN and Cr ≤ 1.5 × ULN; 3) Cardiac ultrasound: Left ventricular ejection fraction (LVEF) ≥ 50%; 11. The subjects voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Individuals with a known history of allergies to the components of this medication regimen;
2. Have other malignant tumors within the past 5 years prior to signing the informed consent form (excluding non melanoma skin cancer or other tumors that have been effectively treated, and malignant tumors that are considered cured);
3. Existence of brain metastases and/or cancerous meningitis;
4. Previously received allogeneic stem cell or parenchymal organ transplantation;
5. Past or current congenital or acquired immunodeficiency diseases;
6. Patients who are known or suspected to have a history of allergies to vediximab or paclitaxel like drugs, or who have a history of hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins, or who are allergic to excipients of the study drug;
7. Other significant clinical and laboratory abnormalities, which the researchers believe will affect the safety evaluation, such as uncontrollable diabetes, hypertension, cirrhosis, interstitial pneumonia, obstructive pulmonary disease, chronic kidney disease, peripheral neuropathy of grade II or above (CTCAE V5.0), thyroid dysfunction, heart failure of NYHA grade 3 or above, etc;
8. Severe infections that are active or poorly controlled clinically; Active infections, including:

   1. AIDS virus (HIV/2 antibody) positive;
   2. Active hepatitis B (HBsAg positive or HBV DNA>2000IU/ml with abnormal liver function);
   3. Active hepatitis C (HCV antibody positive or HCV RNA ≥ 103 copies/ml with abnormal liver function);
   4. Active tuberculosis;
   5. Other uncontrollable active infections (CTCAE V5.0>grade 2);
9. Severe heart disease or discomfort that cannot be treated;
10. Suffering from mental illness or substance abuse, unable to cooperate;
11. Simultaneously participating in other clinical trials;
12. The researchers believe that it is not suitable for the participants to be included.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Prostate Specific Antigen (PSA) ≥50% Response Rate (PSA50) | From treatment administration up to a maximum duration of 36 months
  Will assess PSA decline of ≥50% from baseline (PSA50), using the Prostate Cancer Working Group 3 (PCWG3) criteria.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 3 years
  Objective Response Rate (ORR) assessed according to the evaluation criteria for the efficacy of solid tumors (RECIST v1.1).
Progression Free Survival(PFS) | From treatment administration up to a maximum duration of 36 months
  The time from the beginning of the patient's treatment to the disease progression or death for any reason.Based on RECIST criteria v1.1
Overall Survival(OS) | From treatment administration up to a maximum duration of 36 months
  Time from start of treatment to death due to any cause.
Percentage of Participants With Adverse Events (AEs) | Up to approximately 3 years
  Number of participants with adverse effects of treatment. Frequency and severity of adverse effects of treatment as assessed by NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No